CLINICAL TRIAL: NCT06817382
Title: A Phase 1, Multicenter, Open-label Study to Investigate the Safety and Biodistribution of a Single Intrathecal Injection of INS1201 in Ambulatory Males With Duchenne Muscular Dystrophy (The ASCEND Study)
Brief Title: A Study to Investigate the Safety and Biodistribution of a Single Intrathecal (IT) Injection of INS1201 in Ambulatory Males With Duchenne Muscular Dystrophy (DMD)
Acronym: ASCEND
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Gene Therapy LLC (Industry)
Responsible Party: Sponsor
Organization: Insmed Incorporated (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INS1201-101
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Cohort 1 (Experimental): Participants aged 3 to <5 years will receive a single dose level 1 of INS1201 by IT injection on Day 1.
  Interventions: Genetic: INS1201
- Part 1: Cohort 2 (Experimental): Participants aged 3 to <5 years will receive a single dose level 2 of INS1201 by IT injection on Day 1.
  Interventions: Genetic: INS1201
- Part 2: Cohort 3 (Experimental): Participants aged 2 to <3 years will receive a single dose level 1 of INS1201 by IT injection on Day 1.
  Interventions: Genetic: INS1201
- Part 2: Cohort 4 (Experimental): Participants aged 2 to <3 years will receive a single dose level 2 of INS1201 by IT injection on Day 1.
  Interventions: Genetic: INS1201

INTERVENTIONS:
Genetic: INS1201 — Suspension for IT injection.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a single dose of INS1201 via IT administration in ambulatory male participants with DMD.

ELIGIBILITY:
Inclusion Criteria

* Participant must be male at birth, 3 to <5 years of age, inclusive (Part 1) and 2 to <3 years of age (Part 2), at the time of legally authorized representative (LAR) signing and dating the informed consent form.
* Ambulatory -as defined as the ability to walk at least 10 meters unassisted (ie, without personal assistance or use of any assistive devices) Note: children who have not yet developed the ability to walk by the time of screening (for whatever reason) will not be eligible for the study.
* Has a definitive diagnosis of DMD prior to Screening or as part of Screening based on genetic testing. Note that participants who rescreen do not have to repeat genetic testing for the diagnosis of DMD if one is already on file. Genetic reports must describe a frameshift deletion, frameshift duplication, premature stop ("nonsense"), canonical splice site mutation, or other pathogenic variant in the DMD gene fully contained between exons 18 to 58 (inclusive) that is expected to lead to absence of a functional dystrophin protein (mutations in exons 1-17 or 59-71 are therefore not permitted).
* Able to cooperate with motor assessment testing.
* Has received vaccinations recommended for the participant's age and DMD disease according to Centers for Disease Control and Prevention (CDC) Child and Adolescent Immunization Schedule by Age, World Health Organization, or local recommendation incorporating the Advisory Committee on Immunization Practices (ACIP) Vaccine Recommendations and Guidelines for Patients with Altered Immunocompetence.

Exception is made for seasonal influenza and coronavirus disease 2019 (COVID-19) vaccines, for which shared decision-making with the participant's physician is encouraged.

Exclusion Criteria

* Prior treatment with gene or cell-based therapy at any time.
* Oligonucleotide-based exon skipping or small molecule stop codon readthrough-promoting therapies for at least 6 months prior to enrolment.
* Has left ventricular ejection fraction < 50% on the screening echocardiogram (ECHO) or clinical signs and/or symptoms of cardiomyopathy.
* Has cardiac arrhythmia or significant electrocardiogram (ECG) interval abnormalities.
* Major surgery within 3 months prior to Day 1 or planned surgery or procedures that would interfere with the conduct of the study at any time during this study.
* The presence of any other clinically significant illness, including cardiac, pulmonary, hepatic, renal, hematologic, immunologic/allergic, behavioural disease, infection, unhealed injury, malignancy, concomitant illness, extenuating circumstance, or requirement for chronic drug treatment that, in the opinion of the Investigator:

  1. Creates unnecessary risks for undergoing gene transfer;
  2. Might compromise the participant's ability to comply with the protocol-required testing or procedures; or
  3. Might compromise the participant's well-being, safety, or clinical interpretability.
* Has serological evidence of current, chronic, or active human immunodeficiency virus, hepatitis C, or hepatitis B infection.
* Has signs of clinically significant symptomatic infection (eg, upper respiratory tract infection, pneumonia, pyelonephritis, meningitis) within 4 weeks prior to Day 1.
* Has contraindications for IT administration of the product or for lumbar puncture, such as anatomical abnormalities, bleeding disorders or other medical conditions (eg, spina bifida, meningitis, or significant clotting abnormalities).
* Demonstrates cognitive or developmental delay or impairment that could confound assessment of motor development in the opinion of the Investigator.
* Total serum anti-AAV9 antibody titers of > 1:50 as determined by ELISA within 14 days of Day 1.

Note: Other inclusion/exclusion criteria may apply.

Ages: 2 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Up to Week 96

SECONDARY OUTCOMES:
Parts 1 and 2: Recommended Phase 2 Dose (RP2D) of INS1201 | Week 16
Parts 1 and 2: Change From Baseline in Quantity of Micro-Dystrophin Deoxyribonucleic Acid (DNA) as Measured by Droplet Digital Polymerase Chain Reaction (ddPCR) at Weeks 16 and 48 | Baseline, Weeks 16 and 48
Parts 1 and 2: Change From Baseline in Micro-Dystrophin Protein Expression as Measured by Quantitative Protein Analysis at Weeks 16 and 48 | Baseline, Weeks 16 and 48

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - USA012, Little Rock, Arkansas
  - USA010, Davis, California
  - USA002, Palo Alto, California
  - USA005, San Diego, California
  - Rare Disease Research (USA004), Atlanta, Georgia
  - USA008, Rochester, New York
  - USA006, Columbus, Ohio
  - USA001, Memphis, Tennessee
  - USA015, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No